CLINICAL TRIAL: NCT06820268
Title: A Phase I Trial to Evaluate the Tolerability, Pharmacokinetics and Preliminary Efficacy of XS-04 in Patients with Hematologic Malignancies
Brief Title: A Study of XS-04 in Patients with Relapsed or Refractory Hematologic Malignancies
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: NovaOnco Therapeutics Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XS-04-I101
Record Dates: First submitted 2025-01-09; First posted 2025-02-11 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: B-cell Lymphoma; Acute Myeloid Leukemia; Myelodysplastic Syndrome
MeSH Terms: conditions — Lymphoma, B-Cell; Leukemia, Myeloid, Acute; Myelodysplastic Syndromes

STUDY DESIGN:
Intervention Model Description: A multicenter, open-label, single-arm Phase I dose-escalation and dose-expansion clinical study
Masking Description: Open label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- A multicenter, open-label, single-arm Phase I dose-escalation and dose-expansion clinical study (Experimental): For drugs, use the generic name and include dosage form, dosage, frequency, and duration. Note: Group description not yet entered.] XS-04 tablet specifications: 0.5 mg, 5 mg, 20 mg. Dose escalation phase: 1 mg, 3 mg, 10 mg, 20 mg, 40 mg, 80 mg, 120 mg, 160 mg/day (dose adjustment allowed based on actual escalation situation); Cycle 0 phase, oral administration once (dose is half of the total daily dose for the respective dose group), observe for two days (based on the PK results of the first 1-2 dose groups, decide whether the remaining dose groups need Cycle 0 phase); thereafter Cycle 1-N phase, each 28 days is one treatment cycle, continuous administration, two times daily. Dose regimen adjustments are allowed based on PK, safety, and efficacy data in this trial.
  Dose expansion phase: Based on the results of the dose escalation phase, cohort one and cohort two are planned to use the RP2D dose, cohort three safety lead-in phase is
  Interventions: Drug: XS-04 tablet

INTERVENTIONS:
Drug: XS-04 tablet — Each treatment cycle is 28 days, with continuous oral administration, twice daily.

SUMMARY:
Evaluation of the safety, tolerability, pharmacokinetics, and preliminary efficacy of XS-04 in patients with relapsed or refractory hematologic malignancies

DETAILED DESCRIPTION:
Main Objective: To evaluate the safety and tolerability of XS-04 tablets in patients with relapsed or refractory hematologic malignancies. To determine the maximal tolerated dose (MTD) and/or the recommended phase 2 dose (RP2D) of XS-04 tablets. Secondary Objective: To determine the pharmacokinetic (PK) characteristics of XS-04 tablets after single and multiple oral administrations. To preliminarily evaluate the efficacy of XS-04 tablets in patients with relapsed or refractory hematologic malignancies. Exploratory Objective: To preliminarily assess the metabolic transformation characteristics after oral administration of XS-04 tablets. To evaluate the population PK and exposure-effect (E-R) relationship. To explore the association between relevant biomarkers and drug efficacy; to explore the correlation between PD biomarkers and PK. To assess the impact of food on the PK characteristics of orally administered XS-04 tablets in patients.

ELIGIBILITY:
Inclusion Criteria

Patients must meet all of the following conditions to be enrolled:

* Voluntarily participate in the clinical trial and sign the informed consent form (ICF).
* Age ≥18 years, ≤75 years, regardless of gender.
* Dose escalation phase: Patients with mature B-cell malignant tumors confirmed by histopathology according to the 2017 World Health Organization (WHO) classification, who have failed existing treatments and have no suitable treatment options and have treatment indications.

Dose expansion phase: Patients with B-cell lymphoma confirmed by histopathology according to the 2017 WHO classification (cohort 1 includes DLBCL patients, cohort 2 includes other B-cell lymphoma patients), and patients with myeloid tumors confirmed according to the 2016 WHO classification (cohort 3 includes AML, MDS patients).

Meet the following disease-specific criteria (tumor types not listed below will be discussed by the sponsor and the investigators to decide if they can be enrolled):

1. For indolent B-NHL (follicular lymphoma [FL], marginal zone lymphoma [MZL], and Waldenström macroglobulinemia [WM]), patients must have received at least two lines of systemic therapy, including at least one line of combination therapy containing anti-CD20 antibodies; for chronic lymphocytic leukemia/small lymphocytic lymphoma (CLL/SLL), patients must have received at least two lines of systemic therapy, including BTK inhibitors or BCL-2 inhibitors; for MCL, patients must have received at least two lines of systemic therapy (including anti-CD20 antibodies, BTK inhibitors, etc.); for aggressive B-NHL (DLBCL), patients must have failed or relapsed after at least two lines of systemic therapy and are not suitable for hematopoietic stem cell transplantation.
2. For AML, diagnosed according to the 2016 World Health Organization (WHO) classification, meeting the definition of relapsed/refractory as per the "Chinese Guidelines for the Diagnosis and Treatment of Relapsed/Refractory Acute Myeloid Leukemia (2021 Edition)";
3. For MDS, pathologically confirmed MDS meeting the WHO 2016 classification criteria; and prognostic scoring system assessment as intermediate to high risk (IPSS-R score >3), relapsed or refractory;

   * B-cell lymphoma patients must have at least one radiographically measurable lesion (i.e., lymph node with long diameter [LDi] >1.5 cm, extranodal lesion with LDi >1.0 cm).
   * Patients must be willing to undergo bone marrow aspiration and/or bone marrow biopsy.
   * ECOG score of 0-1 for dose escalation phase; 0-2 for dose expansion phase.
   * Expected survival time ≥3 months.
   * For mature B-cell malignant tumors, during the screening period, there must be sufficient bone marrow not dependent on growth factor support, according to local laboratory reference ranges, as follows:

a. Absolute neutrophil count (ANC) ≥1.0×10^9/L (patients with neutrophils <1.0×10^9/L due to lymphoma bone marrow infiltration may be enrolled at the investigator's discretion); b. Platelets ≥75×10^9/L (dose escalation phase), platelets ≥50×10^9/L (dose expansion phase), no transfusion within 14 days before the first dose; c. Hemoglobin ≥80 g/L. For AML, white blood cell count (WBC) must be ≤20×10^9/L (hydroxycarbamide treatment to reduce white blood cells is allowed).

* Adequate organ function, with laboratory tests within the following requirements within 7 days before the first dose:

  1. Liver function: Serum aspartate aminotransferase (AST), alanine aminotransferase (ALT) ≤2.5×ULN, total bilirubin ≤1.5×upper limit of normal (ULN); if there is liver involvement, AST, ALT ≤5×ULN; total bilirubin ≤3×ULN;
  2. Kidney function: Serum creatinine ≤1.5×ULN or estimated creatinine clearance ≥50 mL/min according to the Cockcroft-Gault formula;
  3. Coagulation function: International normalized ratio (INR) or prothrombin time (PT) ≤1.5×ULN; activated partial thromboplastin time (aPTT) ≤1.5×ULN.
* Female patients of childbearing potential must have a negative serum pregnancy test within 7 days before the first dose during the screening period. Patients must agree to use reliable contraception methods from signing the informed consent form to 3 months after the last dose. These include but are not limited to: abstinence, male vasectomy, female sterilization surgery, effective intrauterine contraceptive device, effective contraceptive drugs.
* Patients must be able to comply with study procedures and protocol-specified visits.

Exclusion Criteria

Patients meeting any of the following conditions are not eligible for this clinical study:

* Burkitt lymphoma/leukemia, plasma cell myeloma, plasmablastic lymphoma.
* Acute promyelocytic leukemia (APL) or BCR-ABL positive AML patients or those with a history of myeloproliferative neoplasms (MPN).
* Use of other cytotoxic drugs, investigational drugs, or other antitumor drugs within 14 days or 5 half-lives before the first dose of the study drug (whichever is shorter) (except hydroxycarbamide and leukapheresis). Patients who received tumor immunotherapy, antibody, or peptide antitumor drug treatment within 4 weeks before the first dose of the study drug.
* Patients who underwent therapeutic surgery other than diagnostic, biopsy, or drainage procedures within 4 weeks before the first dose of the study drug, or who are expected to undergo major surgery during the study. For patients who underwent drainage procedures (e.g., thoracic, biliary, etc.) and/or placement of drainage tubes within 4 weeks before the study drug, related symptoms/signs must have substantially resolved, and no prophylactic/therapeutic use of antibiotics is required.
* Systemic radiotherapy within 4 weeks before the first dose of the study drug.
* Unresolved toxic reactions from previous antitumor treatments (> NCI-CTCAE 5.0 grade 1), alopecia, pigmentation, neurotoxicity, or other toxicities assessed by the investigator as chronic and not affecting the safety of the study drug, resolved to NCI-CTCAE 5.0 grade 2 or below are allowed for enrollment.
* Previous allogeneic stem cell transplantation; autologous stem cell transplantation or adoptive immune cell therapy within 3 months before the first dose of the study drug (mature B-cell malignant tumor patients) or within 6 months (AML, MDS patients).
* Patients with lymphoma/leukemia involving the central nervous system (CNS).
* Dysphagia, or a history of severe gastrointestinal disease (e.g., active inflammatory bowel disease, gastrointestinal perforation) with symptoms that cannot be reasonably controlled; or gastrointestinal diseases affecting drug absorption (e.g., Crohn's disease, ulcerative colitis, ileus, short bowel syndrome) or other malabsorption conditions.
* Patients with ocular conjunctival, corneal lesions (can be enrolled after treatment of ocular lesions is cured).
* Patients with active or unstable cardiovascular and cerebrovascular diseases, including but not limited to:

  1. Severe cardiac rhythm or conduction abnormalities requiring clinical intervention;
  2. Acute coronary syndrome, congestive heart failure, myocardial infarction, unstable angina, coronary/peripheral artery bypass grafting, cerebral infarction, cerebral hemorrhage, pulmonary embolism, deep vein thrombosis (within 3 months before the first dose) or other severe cardiovascular events within 6 months before the first dose;
  3. New York Heart Association (NYHA) heart function classification ≥II;
  4. Left ventricular ejection fraction (LVEF) <50%;
  5. Presence of torsades de pointes, congenital long QT syndrome;
  6. QTcF >450ms (male) or >470ms (female);
  7. Uncontrolled hypertension despite optimal treatment (defined as systolic blood pressure ≥160 mmHg or diastolic blood pressure ≥100 mmHg under medication control).
* History of interstitial lung disease (ILD), pulmonary interstitial fibrosis; or evidence of active pneumonia on chest CT scan during the screening period.
* Patients with congenital immune deficiency diseases, or active autoimmune diseases, including but not limited to active and uncontrolled autoimmune cytopenia, persisting for 2 weeks or longer, including autoimmune hemolytic anemia and idiopathic thrombocytopenic purpura.
* Patients with coagulopathy (e.g., hemophilia).
* Currently using anticoagulant drugs.
* History of severe allergies, or allergies to any active or inactive components of the study drug.
* Uncontrolled systemic infection (viral, bacterial, fungal) within two weeks before the first dose of the study drug; hepatitis B surface antigen positive and hepatitis B virus DNA exceeding 1000 IU/ml; hepatitis C virus (HCV) antibody positive or HCV RNA positive; human immunodeficiency virus (HIV) antibody positive.
* Patients with other primary malignant neoplasms, the following conditions can be enrolled: cured and completely excised basal cell and squamous cell skin cancer, completely excised carcinoma in situ of any type.
* Need to continue using systemic immunosuppressants or systemic corticosteroids (≥10mg prednisone or equivalent of other corticosteroids) within two weeks before the study drug.
* Use of strong CYP3A inhibitors or inducers within two weeks before the first dose.
* Pregnant or lactating women.
* Any other severe or uncontrolled acute or chronic disease or laboratory test abnormality or other reasons deemed unsuitable for participation in this clinical study by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Estimated)
Dates: Start 2025-01-14 (Actual); Primary Completion 2027-11-01 (Estimated); Study Completion 2028-03-15 (Estimated)

PRIMARY OUTCOMES:
The occurrence of treatment-related adverse events meeting the criteria for dose limiting toxicities (DLTs) | At the end of C1D21(each cycle is 28 days)
  Safety indicators
Maximum Tolerated Dose (MTD) and/or Recommended Phase II Dose (RP2D) | Up to 24 months
  Safety indicators and efficacy indicators

SECONDARY OUTCOMES:
The occurrence of adverse events (AEs) reported in all subjects who received study drug | From enrollment up to 30 days after last dose
  Safety indicators
The occurrence of treatment-emergent adverse events (TEAs) | From first dose up to 30 days after last dose
  Safety indicators
Pharmacokinetic variables including maximum plasma concentration (Cmax) | Cycle1(28days）
  Safety indicators
Pharmacokinetic variables including maximum plasma concentration (Cmin) | Cycle1(28days）
  Safety indicators
PK Parameters After Single and Multiple Oral Doses of XS-04 Tablets | Cycle 0 to Cycle 3
  Safety indicators

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - Beijing Cancer Hospital, Beijing
  - Sun Yat-sen University Cancer Center, Guangdong
  - Affiliated Hospital of Hebei University, Hebei
  - Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Hubei

IPD SHARING:
Plan to Share IPD: No